CLINICAL TRIAL: NCT06701344
Title: A Prospective, Multicenter, Single-arm Phase II Clinical Trial to Evaluate the Safety and Efficacy of the Combination Therapy of Go-CHOP in de Novo Intestinal T-cell Lymphoma Patients
Brief Title: Go-CHOP in de Novo Intestinal T-cell Lymphoma Patients
Acronym: GOAL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor and Director，Shanghai Institute of Hematology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOAL
Record Dates: First submitted 2024-11-21; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Enteropathy Associated T Cell Lymphoma
Keywords: Enteropathy-Associated T-Cell Lymphoma; Golidocitinib
MeSH Terms: conditions — Enteropathy-Associated T-Cell Lymphoma | interventions — Cyclophosphamide; Vincristine; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Go-CHOP (Experimental): Golidocitinib 150mg qd plus Standard CHOP regimen
  Interventions: Drug: Go-CHOP (Golidocitinib plus Cyclophosphamide, vincristine, doxorubicin and prednisone); Drug: Golidocitinib

INTERVENTIONS:
Drug: Go-CHOP (Golidocitinib plus Cyclophosphamide, vincristine, doxorubicin and prednisone) — Induction Treatment:
  Golidocitinib:150mg QD Cyclophosphamide:750mg/m2，d1 vincristine:1.4mg/m2，d1(max 2mg) doxorubicin:50mg/m2，d1 Prednisone:60mg/m2 (max 100mg)，d1-d5 Every 21 days
Drug: Golidocitinib — Maintenance Treatment:
  Complete remission patients will further divide into two groups. Unfit, frail old patients will receieve Golidocitinib 150mg QD for two years. Fit, young patients will receive ASCT.

SUMMARY:
The goal of this observational study is to evaluate the safety and efficacy of Go-CHOP (Golidocitinib plus Cyclophosphamide, Hydroxydoxorubicin, Oncovin and Prednisone) in de novo intestinal T-cell lymphoma patients, The aim is to evaluate the complete response rate (CRR). Participants will receive Go-CHOP for 6 cycles every 21 days followed by either maintenance therapy or ASCT.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-75 years old, both male and female participants are eligible; Histopathologically confirmed, untreated intestinal T-cell lymphoma, including: enteropathy-associated T-cell lymphoma, monomorphic epitheliotropic intestinal T-cell lymphoma, intestinal T-cell lymphoma not otherwise specified (NOS), and other subtypes of intestinal T-cell lymphoma deemed appropriate for inclusion by the investigator; Expected survival of ≥12 weeks, with cardiac, pulmonary, hepatic, and renal functions assessed by the investigator as adequate for the proposed treatment regimen; Female participants of childbearing potential and male participants with partners of childbearing potential must agree to and adhere to effective contraceptive measures during the treatment period and for 180 days after the last dose of the study drug; Participants must voluntarily join the study, sign the informed consent form, demonstrate good compliance, and cooperate with follow-up assessments.

Exclusion Criteria:

Involvement of the central nervous system (CNS); Receipt of any antitumor treatment (including radiotherapy, chemotherapy, immunotherapy, targeted therapy, or investigational drugs) within 28 days prior to the first dose or within five half-lives of the antitumor drug, whichever is shorter; Major surgery within 28 days prior to the first dose or planned surgery during the study period; Presence of other uncontrolled malignancies. Early-stage cancers that have been treated with curative intent, such as in situ lung cancer, non-melanoma skin cancers (basal or squamous cell carcinoma), or cervical carcinoma in situ, may be excluded at the investigator's discretion; History of allogeneic hematopoietic stem cell transplantation;

Any of the following treatment histories:

1. Current use (or inability to discontinue use) of strong CYP3A inducers (within at least 3 weeks) or strong inhibitors (within at least 1 week) prior to the first dose;
2. Prior use of JAK or STAT3 inhibitors;
3. Current use of vitamin K antagonists, antiplatelet agents, or anticoagulants (or inability to discontinue these medications within 1 week prior to the first dose);
4. Vaccination with live vaccines within 28 days prior to the first dose (except for attenuated influenza vaccines);

Active infections, including:

1. Known active or latent tuberculosis, including positive tuberculin skin tests (PPD), or findings of active or latent tuberculosis on chest X-ray/CT scans (positive skin test defined as an induration diameter >10 mm or according to local clinical standards);
2. Known history of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome (AIDS);
3. Active chronic hepatitis B or hepatitis C infections, defined as hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody positivity. Patients with HBsAg-negative but hepatitis B core antibody (HBcAb)-positive results must undergo hepatitis B virus DNA testing, and those with HBV DNA ≥1000 IU/mL will be excluded;
4. Active infections requiring treatment within 14 days, including pneumonia;

Poorly controlled cardiac symptoms or diseases, such as:

1. NYHA class > II heart failure;
2. Unstable angina;
3. Myocardial infarction within 1 year;
4. Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
5. Left ventricular ejection fraction (LVEF) ≤ 50%;

Abnormal laboratory test results during screening (unless attributed to lymphoma):

Neutrophils <1.5×10⁹/L; Platelets <75×10⁹/L; ALT or AST >2× upper limit of normal (ULN), alkaline phosphatase (AKP), or bilirubin >1.5× ULN; Creatinine >1.5× ULN; History of interstitial lung disease, excluding asymptomatic, radiation-induced interstitial lung disease; Unresolved drug-related adverse events ≥ grade 2 (CTCAE) prior to the first dose, except for alopecia; Hypersensitivity to golisitinib, capsule excipients, or chemically related compounds; Pregnancy, lactation, or unwillingness to use contraception for female participants of childbearing potential; Known history of substance or drug abuse; Presence of other severe physical or mental illnesses or laboratory abnormalities that may increase study participation risk, interfere with study outcomes, or, in the investigator's opinion, make the patient unsuitable for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-12-04 (Estimated); Primary Completion 2026-05-04 (Estimated); Study Completion 2027-12-04 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | At the end of Cycle 6 (each cycle is 21days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Progression-free survival | Baseline up to data cut-off(up to approximately 3 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Objective Response Rate | At the end of Cycle 6 (each cycle is 21days)
  Percentage of participants with complete or partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Duration of Response | Baseline up to data cut-off(up to approximately 3 years)
  Applicable to complete or partial response participants. DoR was defined as the time from the first documented date of complete or partial response until the date of the disease progression or death from any causes.
Overall survival | Baseline up to data cut-off(up to approximately 3 years)
  Percentage of participants with complete or partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Adverse Events | Baseline up to data cut-off(up to approximately 3 years)
  Adverse Events are assessed based on CTCAE v5.0

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao C, Feng J, Gu H, Tang H, Xu L, Dong H, Dong B, Shu M, Bai Q, Liang R, Zhang T, Yang L, Wang Z, Chen X, Gao G. Distribution of lymphoid neoplasms in Northwest China: Analysis of 3244 cases according to WHO classification in a single institution. Ann Diagn Pathol. 2018 Jun;34:60-65. doi: 10.1016/j.anndiagpath.2017.05.005. Epub 2017 May 12. PMID 29661730
- [Background] Greenplate A, Wang K, Tripathi RM, Palma N, Ali SM, Stephens PJ, Miller VA, Shyr Y, Guo Y, Reddy NM, Kozhaya L, Unutmaz D, Chen X, Irish JM, Dave UP. Genomic Profiling of T-Cell Neoplasms Reveals Frequent JAK1 and JAK3 Mutations With Clonal Evasion From Targeted Therapies. JCO Precis Oncol. 2018;2018:PO.17.00019. doi: 10.1200/PO.17.00019. Epub 2018 Feb 13. PMID 30079384
- [Background] Vose J, Armitage J, Weisenburger D; International T-Cell Lymphoma Project. International peripheral T-cell and natural killer/T-cell lymphoma study: pathology findings and clinical outcomes. J Clin Oncol. 2008 Sep 1;26(25):4124-30. doi: 10.1200/JCO.2008.16.4558. Epub 2008 Jul 14. PMID 18626005
- [Background] d'Amore F, Relander T, Lauritzsen GF, Jantunen E, Hagberg H, Anderson H, Holte H, Osterborg A, Merup M, Brown P, Kuittinen O, Erlanson M, Ostenstad B, Fagerli UM, Gadeberg OV, Sundstrom C, Delabie J, Ralfkiaer E, Vornanen M, Toldbod HE. Up-front autologous stem-cell transplantation in peripheral T-cell lymphoma: NLG-T-01. J Clin Oncol. 2012 Sep 1;30(25):3093-9. doi: 10.1200/JCO.2011.40.2719. Epub 2012 Jul 30. PMID 22851556
- [Background] Malamut G, Chandesris O, Verkarre V, Meresse B, Callens C, Macintyre E, Bouhnik Y, Gornet JM, Allez M, Jian R, Berger A, Chatellier G, Brousse N, Hermine O, Cerf-Bensussan N, Cellier C. Enteropathy associated T cell lymphoma in celiac disease: a large retrospective study. Dig Liver Dis. 2013 May;45(5):377-84. doi: 10.1016/j.dld.2012.12.001. Epub 2013 Jan 10. PMID 23313469
- [Background] Sharaiha RZ, Lebwohl B, Reimers L, Bhagat G, Green PH, Neugut AI. Increasing incidence of enteropathy-associated T-cell lymphoma in the United States, 1973-2008. Cancer. 2012 Aug 1;118(15):3786-92. doi: 10.1002/cncr.26700. Epub 2011 Dec 13. PMID 22169928
- [Background] West J, Jepsen P, Card TR, Crooks CJ, Bishton M. Incidence and Survival in Patients With Enteropathy-associated T-Cell Lymphoma: Nationwide Registry Studies From England and Denmark. Gastroenterology. 2023 Oct;165(4):1064-1066.e3. doi: 10.1053/j.gastro.2023.06.003. Epub 2023 Jun 9. No abstract available. PMID 37301328
- [Background] Verbeek WH, Van De Water JM, Al-Toma A, Oudejans JJ, Mulder CJ, Coupe VM. Incidence of enteropathy--associated T-cell lymphoma: a nation-wide study of a population-based registry in The Netherlands. Scand J Gastroenterol. 2008;43(11):1322-8. doi: 10.1080/00365520802240222. PMID 18618372
- [Background] Al-Toma A, Goerres MS, Meijer JW, Pena AS, Crusius JB, Mulder CJ. Human leukocyte antigen-DQ2 homozygosity and the development of refractory celiac disease and enteropathy-associated T-cell lymphoma. Clin Gastroenterol Hepatol. 2006 Mar;4(3):315-9. doi: 10.1016/j.cgh.2005.12.011. PMID 16527694
- [Background] Sieniawski M, Angamuthu N, Boyd K, Chasty R, Davies J, Forsyth P, Jack F, Lyons S, Mounter P, Revell P, Proctor SJ, Lennard AL. Evaluation of enteropathy-associated T-cell lymphoma comparing standard therapies with a novel regimen including autologous stem cell transplantation. Blood. 2010 May 6;115(18):3664-70. doi: 10.1182/blood-2009-07-231324. Epub 2010 Mar 2. PMID 20197551
- [Background] Gale J, Simmonds PD, Mead GM, Sweetenham JW, Wright DH. Enteropathy-type intestinal T-cell lymphoma: clinical features and treatment of 31 patients in a single center. J Clin Oncol. 2000 Feb;18(4):795-803. doi: 10.1200/JCO.2000.18.4.795. PMID 10673521
- [Background] Delabie J, Holte H, Vose JM, Ullrich F, Jaffe ES, Savage KJ, Connors JM, Rimsza L, Harris NL, Muller-Hermelink K, Rudiger T, Coiffier B, Gascoyne RD, Berger F, Tobinai K, Au WY, Liang R, Montserrat E, Hochberg EP, Pileri S, Federico M, Nathwani B, Armitage JO, Weisenburger DD. Enteropathy-associated T-cell lymphoma: clinical and histological findings from the international peripheral T-cell lymphoma project. Blood. 2011 Jul 7;118(1):148-55. doi: 10.1182/blood-2011-02-335216. Epub 2011 May 12. PMID 21566094